CLINICAL TRIAL: NCT01500694
Title: A Phase 3, Open-label, Multicentre Study to Provide Access to Guanfacine Hydrochloride Extended-release for European Subjects With Attention-deficit/Hyperactivity Disorder (ADHD) Who Participated in Study SPD503-315 or SPD503-316
Brief Title: Access to Extended Release Guanfacine HCl for Subjects Who Participated in Studies SPD503-315 or SPD503-316 in Europe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD503-318; 2011-004668-31 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extended-release Guanfacine HCl (Experimental)
  Interventions: Drug: Extended-release Guanfacine HCl (Intuniv, SPD503)

INTERVENTIONS:
Drug: Extended-release Guanfacine HCl (Intuniv, SPD503) — Subjects will be dosed orally once-daily in the AM at 1, 2, 3, 4, 5, 6, or 7 mg according to subjects weight and age
  Other Names: Intuniv; SPD503

SUMMARY:
For subjects in Europe that have already participated in either Study SPD503-315 or SPD503-316. This is an extension study that will allow participants access to Extended-release Guanfacine Hydrochloride (HCl) for up to 2 years. This study will help the sponsor evaluate long-term safety and tolerability of Extended-release Guanfacine HCl (SPD503).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects where Study SPD503-318 was not available at the time of their final visit in the antecedent study (SPD503-315 or SPD503-316), may still be screened unless they are well-controlled on another ADHD medication with acceptable tolerability and the parent/caregiver is satisfied with their current ADHD medication.
2. Subject satisfied all entry criteria for the antecedent study (SPD503 315 or SPD503-316).
3. Subject who is a female of child-bearing potential (FOCP), defined as >9 years of age or <9 years of age and is post-menarchal, must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test at the Screening Visit (Visit 1) and a negative urine pregnancy test at the Baseline Visit (Visit 2) and agree to comply with any applicable contraceptive requirements of the protocol.
4. Subject's parent or legally authorised representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations, before completing any study-related procedures.
5. Subject and parent/LAR are willing, able, and likely to fully comply with all the testing and requirements defined in this protocol, including oversight of dosing. Specifically, the parent/LAR must be available upon awakening, to dispense the dose of investigational product for the duration of the study.
6. Subject has a supine and standing blood pressure (BP) measurement within the 95th percentile for age, sex, and height.
7. Subject is functioning at an age-appropriate level intellectually, as deemed by the Investigator.
8. Subject is able to swallow intact tablets.

Exclusion Criteria:

1. Subject has any current, controlled (requiring a prohibited medication or behavioural modification program) or uncontrolled, co-morbid psychiatric diagnosis (except oppositional defiant disorder), including any severe comorbid Axis II disorders or severe Axis I disorders such as post traumatic stress disorder, bipolar illness, psychosis, pervasive developmental disorder, obsessive-compulsive disorder, substance abuse disorder, or other symptomatic manifestations or lifetime history of bipolar illness, psychosis or conduct disorder that, in the opinion of the Investigator, contraindicate treatment with SPD503 or confound efficacy or safety assessments. The Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime version (K-SADS-PL) rating from the antecedent study should be reviewed to confirm diagnosis, if necessary.
2. Subject who early terminated from Study SPD503-315 or Study SPD503-316 for protocol non-adherence, subject non-compliance, an AE, SAE, or withdrawal by subject.
3. Subject experienced any clinically significant AE in their prior SPD503 study (SPD503-315 or SPD503 316) that, in the opinion of the Investigator, would preclude exposure to SPD503.
4. Clinically important abnormality on urine drug and/or alcohol screen at the Screening Visit (Visit 1).
5. Subject has taken any investigational product as follows: last dose of investigational product in Study SPD503-315 within 7 days prior to the Baseline Visit (Visit 2); investigational product in Study SPD503 316 within 30 days prior to the Baseline Visit (Visit 2); any other investigational product within 30 days prior to the Baseline Visit (Visit 2) or any other ADHD medication within 30 days prior to Baseline Visit (Visit 2).
6. Subject is significantly overweight based on Center for Disease Control and Prevention Body Mass Index (BMI)-for-age sex-specific charts at the Screening Visit (Visit 1). Significantly overweight is defined as a BMI >95th percentile.
7. Children aged 6 12 years with a body weight of less than 25.0kg or adolescents aged 13 years and older with a body weight of less than 34.0kg at the Screening Visit (Visit 1).
8. Subject has any condition or illness including clinically significant abnormal laboratory values at the Screening Visit (Visit 1) which, in the opinion of the Investigator, represents an inappropriate risk to the subject and/or could confound the interpretation of the study.
9. Subject is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.
10. Subject has clinically significant ECG findings, as judged by the Investigator with consideration of the central ECG laboratory's interpretation, at the Baseline Visit (Visit 2).
11. Subject has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride, or any components found in SPD503.
12. Subject has a history of alcohol or other substance abuse or dependence, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text RevisionÒ (DSM-IV-TRÒ; with the exception of nicotine) within the last 6 months.
13. Subject has a history of a seizure disorder (other than a single childhood febrile seizure occurring before the age of 3 years) or the presence of a serious tic disorder including Tourette's syndrome.
14. Subject has a known history or presence of structural cardiac abnormalities, serious heart rhythm abnormalities, syncope, cardiac conduction problems (eg, clinically significant heart block), exercise related cardiac events including syncope and pre syncope, or clinically significant bradycardia.
15. Subject with orthostatic hypotension or a known history of controlled or uncontrolled hypertension.
16. Current use of any prohibited medication or other medications, including herbal supplements, that affect BP or heart rate or that have central nervous system (CNS) effects or affect cognitive performance, such as sedating antihistamines and decongestant sympathomimetics (inhaled bronchodilators are permitted) or a history of chronic use of sedating medications (ie, antihistamines) in violation of the protocol specified washout criteria at the Baseline Visit (Visit 2).
17. Subject has a medical condition, other than ADHD, that requires treatment with medications that have CNS effects and/or affect performance.
18. Subject is female and is pregnant or currently lactating.
19. Subject failed screening or was previously enrolled in this study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2012-03-20 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (60):
- Austria (2):
  - Medizinische Universitat Graz Univ fur Kinder, Graz
  - Institut fur Psychosomatik, Vienna
- Belgium (4):
  - Universitaire Kinder-end Jeugdpsychatrie, Hoboken
  - Centre de Reference Neuropediatrique Multidisciplinaire, Namur
  - Huisartspraktijk Jaak Mortelmans, Oostham
  - Zlekenhuis Inkendaal Koninklijke Instelling v.z.w., Vlezenbeek
- France (3):
  - Centre Hospitalier Universitaire Amiens, Amiens, Picardie
  - Centre Hospitalier Charles Perrens, Bordeaux
  - Hopital Gui de Chauliac, Montpellier
- Germany (13):
  - Dr. med. Andreas Mahler, Achim
  - Emovis GmbH, Berlin
  - Sozialpsychitrisches Zentrum, Dorsten
  - Klinik und Poliklinik fur Kinder-und Jugendpsychiatrie un psychotherapie, Dresden
  - Dr. med Walter Robert Otto, Fulda
  - Dr. med. Christian Wolff, Hagen
  - Dr. med Friedrich Kaiser, Hamburg
  - Institut fur Ganzheitliche Medizin und Wissenschaft GmbH, Hüttenberg
  - Friedrich Schiller Universitat Jena Klinik fur Kinder und Jugendpsychiatrie, Jena
  - Universitatsmedizin der Johannes-Gutenberg-Universitat, Mainz
  - Kinder-und Jugendpsychiatrische Praxis, München
  - Somni bene GmbH Institut fur Medizinische Forschung und Schlatmedizin, Schwerin
  - Universitatsklinik Ulm, Ulm
- Our Lady's Children's Hospital, Crumlin, Dublin, Ireland
- Italy (6):
  - Azienda Ospedaliero-Universitaria Policlinico-Vittorio, Catania
  - Azienda Ospedallera G Salvini - Ospedale Di Circolo de RHO, Milan
  - Azienda Ospedallera Fatebenefratelli, Milan
  - U.O di Neuropsichiatria Infantile, Padua
  - IRCCS Fondazione Stella Maris, Pisa
  - Ospedale Policlinico GB Rossi, Verona
- Netherlands (2):
  - Flevo Research, Almere Stad
  - Mondriaan Zorggroep, Heerlen
- Poland (5):
  - NZOZ Gdanskie Centrum Zdrowia, Gdansk
  - Centrum Badari Klinicznych House Sp. z.o.o., Gdansk
  - Gabinet Psychiatrii Doroslych, Dzieci i Mlodziezy, Torun
  - Indywidualna Specjalisyczna Praktyka Lekarska, Torun
  - Contrum Neurospychiatrii Neuromed, Wroclaw
- Romania (3):
  - Spitalul Clinic de Urgenta pentru Copli, Timișoara, Timiș County
  - Spitalul Clinic de Psihiatrie, Bucharest
  - Spitalul Clinic de Psihiatrie Socoia, Iași
- Spain (7):
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitani Vall d'Hebron, Barcelona
  - Hospital Infanta Leonor, Servicio de Psiquiatria, Madrid
  - Hospital Fundacion Alcorcon, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Unidad de Salud Mental Infanto Juvenil, Santander
  - Instituto Valenciano de Neurologia Pediatrica, Valencia
- Drottning Silvias Barnsjukhus, Gothenburg, Sweden
- Ukraine (7):
  - Regional Clinical Psychiatric Hospital, Donetsk
  - Institute of Neurology, Psychiatry and Narcology, Kharkiv
  - Institute of Health Care for Children and Teenagers, Kharkiv
  - Lviv Regional Clinical Psychiatric Hospital, Lviv
  - Odesa Regional Psychoneurological Dispensary, Odesa
  - Poltava Regional Clinical Psychiatric Hospital, Poltava
  - Vinnitsya regional psychoneurological hospital, Vinnytsia
- United Kingdom (6):
  - Lister Hospital, Stevenage, Herfordshire
  - Queen Elizabeth II Hospital - Howlands, Welwyn Garden City, Herfordshire
  - Alder Hey Children's NHS Foundation Trust, West Derby, Liverpool
  - The Children's Centre, Norwich
  - Ryegate Children's Centre, Sheffield
  - Centenary House Child and Adolescent Mental Health Services, Sheffield

REFERENCES:
- [Result] Huss M, Dirks B, Gu J, Robertson B, Newcorn JH, Ramos-Quiroga JA. Long-term safety and efficacy of guanfacine extended release in children and adolescents with ADHD. Eur Child Adolesc Psychiatry. 2018 Oct;27(10):1283-1294. doi: 10.1007/s00787-018-1113-4. Epub 2018 Feb 13. PMID 29442229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 52 sites in 11 countries in Europe: Austria, Belgium, France, Germany, Italy, The Netherlands, Poland, Romania, Spain, Ukraine, and United Kingdom.
Pre-assignment Details: Overall 218 participants screened, of them 215 were enrolled and 214 were treated in the study.The first participant's consent was obtained on 20 March 2012 and last participant assessment took place on 15 September 2015.
Groups:
- SPD503 (6-12 Years): Participants aged 6-12 years received extended-release guanfacine hydrochloride (SPD503) one tablet (1 x 1 milligram [mg] or 2 mg or 3 mg or 4mg) or two tablets (1 x 2+3 mg or 1 x 2+4 mg, 1 x 3+4 mg) once daily for up to 2 years.
- SPD503 (13-18 Years): Participants aged 13-18 years received extended-release guanfacine hydrochloride (SPD503) one tablet (1 x 1 mg or 2 mg or 3 mg or 4mg) or two tablets (1 x 2+3 mg or 1 x 2+4 mg, 1 x 3+4 mg) once daily for up to 2 years.
Period: Overall Study
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Started | 131 | 83 (Participants who received treatment were reported as Started.)
Completed | 79 | 54
Not Completed | 52 | 29
Not completed — Adverse Event | 4 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 23 | 14
Not completed — Lost to Follow-up | 2 | 3
Not completed — Lack of Efficacy | 14 | 5
Not completed — Other | 9 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who took at least 1 dose of SPD503.
Groups:
- SPD503 (6-12 Years): Participants aged 6-12 years received extended-release guanfacine hydrochloride (SPD503) one tablet (1 x 1 mg or 2 mg or 3 mg or 4mg) or two tablets (1 x 2+3 mg or 1 x 2+4 mg, 1 x 3+4 mg) once daily for up to 2 years.
- Total: Total of all reporting groups
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years) | Total
Number analyzed (Participants) | 131 | 83 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (1.56) | 14.7 (1.49) | 11.7 (2.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 105 | 53 | 158

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Systolic Blood Pressure at Final Assessment
Description: Systolic Blood pressure was measured at supine and standing position and mean supine systolic blood pressure was reported here. Final Assessment is the last valid assessment obtained after Baseline (Visit 2/Day 0) whilst on investigational product and before first dose taper medication [Visit 19/Early Termination (ET)/Day 714].
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: Safety Analysis Set includes all enrolled participants who took at least 1 dose of SPD503. Here, n = number of participants analysed for the specific categories for each arm respectively.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 131 | 83
millimeter of mercury (mmHg)
  Baseline (n = 131, 83) | 107.5 (8.73) | 113.5 (9.23)
  Change at Final Assessment (n = 130, 82) | 0.9 (9.35) | 0.3 (9.32)

2. Primary Outcome: Change From Baseline in Mean Diastolic Blood Pressure at Final Assessment
Description: Diastolic Blood pressure was measured at supine and standing position and mean supine diastolic blood pressure was reported here. Final Assessment is the last valid assessment obtained after Baseline (Visit 2/Day 0) whilst on investigational product and before first dose taper medication (Visit 19/ET/Day 714).
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: Safety Analysis Set included all enrolled participants who took at least 1 dose of SPD503. Here, n = number of participants analysed for the specific categories for each arm respectively.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 131 | 83
millimeter of mercury (mmHg)
  Baseline (n=131, 83) | 64.3 (8.12) | 66.8 (9.14)
  Change at Final Assessment (n = 130, 82) | 0.2 (8.96) | 0.1 (9.55)

3. Primary Outcome: Change From Baseline in Mean Supine Pulse at Final Assessment
Description: Pulse was measured at supine and standing position and mean supine pulse was reported here. Final Assessment is the last valid assessment obtained after Baseline (Visit 2/Day 0) whilst on investigational product and before first dose taper medication (Visit 19/ET/Day 714).
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 131 | 83
beats per minute (bpm)
  Baseline (n = 131, 83) | 79.3 (11.17) | 72.1 (9.91)
  Change at Final Assessment (n = 130, 82) | -7.1 (13.52) | -2.9 (11.71)

4. Primary Outcome: Change From Baseline in Mean Height at Final Assessment
Description: Final Assessment is the last valid assessment obtained after Baseline (Visit 2/Day 0) whilst on investigational product and before first dose taper medication (Visit 19/ET/Day 714).
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 131 | 83
centimeter (cm)
  Baseline (n = 131, 83) | 142.03 (10.916) | 166.32 (9.274)
  Change at Final Assessment (n = 128, 79) | 8.80 (5.075) | 5.54 (5.491)

5. Primary Outcome: Change From Baseline in Mean Weight at Final Assessment
Description: as for outcome 4
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 131 | 83
kilogram (kg)
  Baseline (n = 131, 83) | 37.29 (9.256) | 58.53 (11.478)
  Change at Final Assessment (n = 128, 79) | 8.96 (5.886) | 6.74 (5.859)

6. Primary Outcome: Change From Baseline in Electrocardiogram Result (QRS Interval) at Final Assessment
Description: as for outcome 4
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 131 | 83
millisecond (ms)
  Baseline (n=131, 83) | 84.9 (7.72) | 89.7 (6.22)
  Change at Final Assessment (n=127, 77) | 1.8 (6.00) | 1.8 (6.16)

7. Primary Outcome: Change From Baseline in Electrocardiogram Result (QT Interval) at Final Assessment
Description: as for outcome 4
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 131 | 83
millisecond (ms)
  Baseline (n = 131, 83) | 361.4 (21.40) | 375.9 (24.93)
  Change at Final Assessment (n = 127, 77) | 16.9 (27.87) | 9.5 (29.93)

8. Primary Outcome: Number of Participants With Suicidal Behavior and / or Ideation ("Yes" Response) on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a clinician rated assessment of suicidal behavior and / or intent categorized as: Suicidal behavior=a "yes" response to any of 5 suicidal behavior questions (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide); Suicidal ideation=a "yes" response to any one of 5 suicidal ideation questions which includes wish to be dead, and 4 different categories of active suicidal ideation (thought, thought with method, thought with intent, thought with plan and intent).
Time Frame: Final Assessment (last non missing data/up to Day 714)
Population: Safety Analysis Set included all enrolled participants who took at least 1 dose of SPD503 with number of participants evaluable for this outcome at specific categories.
Measure: Number; unit: participants
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 131 | 83
participants
  Suicidal Ideation: Wish to be Dead: number analyzed (Participants) | 130 | 82
  Suicidal Ideation: Wish to be Dead | 0 | 1
  Suicidal Ideation: Non-specific Suicidal Thoughts: number analyzed (Participants) | 130 | 82
  Suicidal Ideation: Non-specific Suicidal Thoughts | 0 | 0
  Suicidal Behaviour: Actual Attempt: number analyzed (Participants) | 130 | 82
  Suicidal Behaviour: Actual Attempt | 0 | 0
  Suicidal Behaviour: Non-Suicidal Self-Injurious: number analyzed (Participants) | 130 | 82
  Suicidal Behaviour: Non-Suicidal Self-Injurious | 0 | 1
  Suicidal Behaviour: Interrupted Attempt: number analyzed (Participants) | 130 | 82
  Suicidal Behaviour: Interrupted Attempt | 0 | 0
  Suicidal Behaviour: Aborted Attempt: number analyzed (Participants) | 130 | 82
  Suicidal Behaviour: Aborted Attempt | 0 | 0

9. Secondary Outcome: Change From Baseline in Attention-deficit and Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) - Total Score at Final Assessment
Description: ADHD-RS-IV was developed to measure the behaviours of children with ADHD with 18 items. Each item is scored from a range of 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items may be grouped into 2 subscales: hyperactivity/impulsivity (even numbered items 2-18) and inattentiveness (odd numbered items 1-17) with possible score range from 0 (no symptoms) to 27 (most severe symptoms). The ADHD-RS-IV possible total scores range from 0 (no symptoms) to 54 (most severe symptoms). Final Assessment is the last valid assessment obtained after Baseline (Visit 2/Day 0) whilst on investigational product and before first dose taper medication (Visit 19/ET/Day 714).
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: Full Analysis Set included enrolled participants who took at least 1 dose of SPD503, excluding participants from site 403. Here, n = number of participants analysed for the specific categories for each arm respectively.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 128 | 81
units on a scale
  Baseline (n = 127, 81) | 40.0 (0.78) | 31.2 (1.19)
  Change at Final Assessment (n = 126, 80) | -20.2 (1.10) | -19.3 (1.31)

10. Secondary Outcome: Number of Participants Assessed With Clinical Global Impression Severity of Illness (CGI-S) Scale
Description: The CGI-S evaluate each participant's severity and improvement over time. The severity of a participant's condition is rated on a 7-point scale ranging from 1 to 7. The scale measures 0 = Not assessed, 1 = Normal, not at all ill, 2 = Borderline mentally ill (BL-MI), 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, 7 = Among the most extremely ill participant. Final Assessment is the last valid assessment obtained after Baseline (Visit 2/Day 0) whilst on investigational product and before first dose taper medication (Visit 19/ET/Day 714).
Time Frame: Baseline (Day 0) and Final Assessment (last non missing data/up to Day 714)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Number analyzed (Participants) | 128 | 81
participants
  Baseline: Normal/BL-MI (n=127,81) | 0 | 2
  Baseline: Mildly ill or greater (n=127, 81) | 127 | 79
  Final assessment: Normal/BL-MI (n=127,80) | 45 | 51
  Final Assessment:Mildly ill or greater(n=127,80) | 82 | 29

ADVERSE EVENTS:
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration (up to Week 105)
Arm/Group | SPD503 (6-12 Years) | SPD503 (13-18 Years)
Serious Adverse Events (participants affected / at risk) | 8/131 | 2/83
Other Adverse Events (participants affected / at risk) | 102/131 | 55/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD503 (6-12 Years) (N=131) | SPD503 (13-18 Years) (N=83)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD503 (6-12 Years) (N=131) | SPD503 (13-18 Years) (N=83)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 8 (11) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (15) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (12) | 3 (4)
Fatigue (General disorders) | 30 (43) | 13 (15)
Pyrexia (General disorders) | 8 (9) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (14) | 18 (24)
Rhinitis (Infections and infestations) | 8 (11) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 9 (16) | 4 (10)
Dizziness (Nervous system disorders) | 12 (16) | 9 (10)
Headache (Nervous system disorders) | 38 (91) | 23 (43)
Somnolence (Nervous system disorders) | 50 (81) | 27 (37)
Aggression (Psychiatric disorders) | 7 (7) | 2 (2)
Insomnia (Psychiatric disorders) | 10 (10) | 6 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.